CLINICAL TRIAL: NCT02098785
Title: Phase I Clinical Trial Investigating the Effects of Caffeine Citrate on Serum Vascular Adhesion Protein -1 (VAP-1) Levels in Healthy Volunteers.
Brief Title: Inhibition of VAP-1 by Caffeine in Healthy Human Volunteers Study
Acronym: NOCTUA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Local resource issue - never actually started post ethics approval.
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RG_14-045
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2017-05

CONDITIONS: Liver Disease
Keywords: VAP; liver; hepatology; caffeine
MeSH Terms: conditions — Liver Diseases | interventions — caffeine citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Caffeine citrate (Peyona) 400mg (Experimental): Caffeine Citrate (Peyona) 400mg single dose (20ml oral solution)
  Interventions: Drug: Caffeine citrate

INTERVENTIONS:
Drug: Caffeine citrate — Oral solution
  Other Names: Peyona

SUMMARY:
Worldwide, liver related morbidity and mortality continue to rise. It is the 5th commonest cause of death in the UK. Liver damage consists of two main components - a) damage to the cells of the liver, called hepatocytes, meaning the liver cannot function properly leading to jaundice (yellow appearance of the skin and/or eyes) and liver failure and b) scarring of the liver, called Cirrhosis, leading to impaired function and inadequate blood flow through the liver with potential to develop into cancer. Manifestations of this state include ascites (fluid in the tummy) and varices (swollen blood vessels in the food pipe). Liver transplant is currently the only curative treatment for end stage chronic liver disease. Unfortunately its high demand has not been matched by an equivalent rise in liver donations and even when a transplant has occurred there are numerous lifestyle effects such as immunosuppression and kidney impairment thus outcome remains poor for many patients. Coffee has been shown to have mortality benefit in humans and drinking two to three cups a day was associated with a 40% reduced risk of developing cirrhosis, particularly alcohol related; and higher the more cups consumed. Previous work has demonstrated coffee reduces the level of fibrosis in the liver by interrupting signalling pathways, blocking the effects of special products, called cytokines, and reducing accumulation of iron. The investigators' hypothesis is that given the potential for caffeine to be used as a treatment in SSAO activity associated diseases it is important to see if the activity of SSAO can be blocked in healthy humans too. The Investigators' aim to examine the effect of caffeine on circulating VAP-1 levels in large numbers of healthy volunteers to assess its potential as an attractive therapeutic target in view of its low toxicity and widespread availability.

DETAILED DESCRIPTION:
One such enzyme known as VAP-1 (vascular adhesion protein-1) is expressed at high levels in liver endothelial cells and studies involving blockage of VAP-1 activity have demonstrated it is involved in a reaction where break down products such as hydrogen peroxide and ammonia active signalling pathways to assist in the movement of cells from blood vessels to the liver. VAP-1 levels become elevated during chronic inflammation in blood vessels of the gut, tonsils, skin and synovium albeit most selectively in liver. Recently, circulating VAP-1 has been demonstrated to be elevated in certain liver diseases particularly alcoholic liver disease. Initial animal studies have shown that activity of the enzyme SSAO (Semicarbazide-sensitive amine oxidase) can be effectively blocked by caffeine administration and that caffeine also blocks the activity of fat cells, known as adipose cells, thus protective against obesity too. SSAO arises from the same family of enzymes as VAP-1 thus importantly shares transferable properties. This information led to small, experimental studies in human liver that corroborate these findings but did not show how caffeine was affecting VAP-1 in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human volunteers aged 18-70 inclusive
* No significant medical problems (as determined by a screening questionnaire)
* Written informed consent given by the patient

Exclusion Criteria:

* Currently pregnant or breast feeding
* Psychiatric, addictive or any disorder which compromises ability to give truly informed consent for participation in this study or comply with the requirements of the study
* Other serious underlying medical conditions that could impair the ability of the patient to participate in the study
* Unable to travel for study visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
VAP-1 serum levels | VAP-1 serum levels at 60, 90 and 120 minutes post administration of caffeine citrate (Peyona)
  The aim of the trial is to examine whether caffeine blocks vascular adhesion protein-1 (VAP-1) activity in the blood of healthy human volunteers and thus prove to be of medicinal value in liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: David Adams, MD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, UK, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided